CLINICAL TRIAL: NCT04651127
Title: Toripalimab, a Anti-PD-1 Antibody, and Histone Deacetylase Inhibitor Chidamide in Patients With Persistent, Recurrent, or Metastatic Cervical Cancer, a Multicenter, Open-label, Single-arm, Phase Ib/II Trial
Brief Title: Anti-PD-1 Antibody Combined With Histone Deacetylase Inhibitor in Patients With Advanced Cervical Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xin Huang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-229-01
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Cervical Cancer; Cervix Cancer; Cervix Neoplasm
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — toripalimab; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab + Chidamide Arm (Experimental)
  Interventions: Drug: Toripalimab + Chidamide

INTERVENTIONS:
Drug: Toripalimab + Chidamide — In combination dose finding phase, phase 1b will begin with Dose Level 1: chidamide 30 mg/day orally (twice a week) and toripalimab (240mg q3w, intravenously) will be administered to eligible subjects on a 21-day treatment cycle. Two dose de-escalation steps are included: Dose Level 2 (chidamide 25 mg/day orally, twice a week and toripalimab 240mg q3w, intravenously) and Dose Level 3 (chidamide 20 mg/day orally, twice a week and toripalimab 240mg q3w, intravenously). If RP2D was reached in Part A, eligible patients would be enrolled and receive toripalimab (240mg q3w, intravenously) plus chidamide (RP2D, twice a week).

SUMMARY:
Cervical cancer is the second-most common cancer in the world and is a leading cause of cancer death among women in developing countries. Cisplatin-based chemotherapy +/- bevacizumab have been recommended as the first-line treatment for patients who present with metastatic (e.g. stage IVB), persistent, or recurrent cervical cancer. However, patients in this setting are rarely curable. Pembrolizumab has been approved for second-line treatment in patients with advanced PD-L1-positive cervical cancer. However, the response rate achieved by PD-1 inhibitors as monotherapy is only modest. Preclinical studies found that in mouse models of B-cell lymphoma, adding a histone deacetylase (HDAC) inhibitor sensitized cancers to anti-PD-1 therapy. Recently, combination treatment of HDAC inhibitors with immune checkpoint inhibitors is widely investigated and has promising results in several cancer types. Toripalimab is a humanized IgG4 monoclonal antibody against PD-1. Chidamide is a class I HDAC inhibitor. Here we conducted a phase Ib/II, single-arm, multi-center study to evaluate the efficacy and safety of toripalimab in combination with chidamide in patients with metastatic, persistent, or recurrent cervical cancer.

DETAILED DESCRIPTION:
There are two main parts to this study; Part A, combination dose finding and Parts B, dose expansion. Part B will either be initiated if RP2D reached in Part A, or not initiated if RP2D was not reached in Part A. Part A has been designed to identify the recommended dose of combination of toripalimab plus chidamide for further clinical evaluation based upon assessment of the safety and tolerability data collected during the first 28 days. "3+3"design was used in the dose finding cohort. If RP2D was reached in Part A, eligible patients would be enrolled and receive toripalimab (240mg q3w, intravenously) plus chidamide (RP2D, twice a week) till disease progression (PD) withdraw of consent, or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF).
2. Patients must have histologically confirmed diagnosis of metastatic, recurrent or persistent squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix which is not amenable to curative treatment with surgery and/or radiation therapy.
3. Age ≥ 18 years and ≤ 70 years.
4. Patients must have measurable disease per RECIST v1.1; measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded as ≥ 10 mm with computed tomography (CT) scan, magnetic resonance imaging (MRI); a lymph node must be ≥ 15 mm in short axis. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy exceeds 3 months.
7. Patients must have progressed on at least one line of platinum-based systemic therapy.

   Note: Prior adjuvant therapy is NOT counted as a systemic chemotherapeutic regimen for management of recurrent, persistent or metastatic cervical cancer. However, adjuvant chemotherapy could be counted as one prior regimen in patients who had recurrence during or within 6 months of completion of therapy.
8. Patients must have adequate organ function as defined by the following criteria:

   * Absolute neutrophil count (ANC) (≥ 1.5×10^9/L), hemoglobin of ≥ 90 g/L, platelets ≥ 80 ×10^9/L
   * Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
   * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 × ULN (however, patients with known liver metastasis who have AST or ALT level ≤ 5 × ULN may be enrolled)
   * Serum creatinine ≤ 1.5 × ULN or creatinine clearance rate ≥ 60 ml/min (Cockcroft-Gault formula)
   * Baseline albumin ≥ 28 g/L
   * Thyroid-stimulating hormone (TSH) levels ≤ 1 × ULN (however, patients with free Triiodothyronine [FT3] or free Thyroxine [FT4] levels ≤ 1 × ULN may be enrolled)

Exclusion Criteria:

1. Prior exposure to immune checkpoint inhibitors, including but not limited to other anti-PD-1 and anti-PD-L1 antibodies, or prior exposure to HDAC inhibitors.
2. Any condition requiring systemic treatment with corticosteroids (>10 mg daily prednisone or equivalents) or other immunosuppressive medications within 14 days before first dose of study drug. Corticosteroids for topical use, nasal spray, and inhaled steroids are allowed.
3. Active autoimmune diseases that require systemic treatment. Alternative treatments (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are permitted.
4. Clinically significant cardiovascular diseases, including but not limited to congestive heart failure (New York heart association [NYHA] class > 2), unstable or severe angina, severe acute myocardial infarction within 1 year before enrollment, supraventricular or ventricular arrhythmia which need medical intervention, or QT interval male ≥ 450 ms, female ≥ 470 ms.
5. Arterial or venous thrombosis within 6 months before enrollment
6. Uncontrolled hypertension defined as systolic pressure ≥ 160 mmHg and/or diastolic pressure ≥ 100 mmHg despite antihypertensive drugs.
7. Proteinuria ≥ (++) or 24 hours total urine protein > 1.0 g.
8. Coagulation abnormalities (INR > 2.0, PT > 16s), with bleeding tendency or are receiving thrombolytic or anticoagulant therapy.
9. Has known active central nervous system metastases.
10. Patients had a diagnosed and/or treated additional malignancy within the last 5 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
11. Has a known history of immunodeficiency including human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease.
12. Has known active Hepatitis B or Hepatitis C.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of the combination of toripalimab and chidamide (Phase Ib) | first 28 days of treatment
  Dose-limiting toxicities (DLTs) are defined as: grade 3 febrile neutropenia, grade 4 hematologic toxicities, and grade 3 non-hematologic toxicities according to CTCAE v5.0
Objective Response Rate (ORR) (Phase II) | from the first drug administration up to two years
  ORR is the proportion of patients with best response of complete response (CR) and partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | from the first drug administration up to two years
  Time from the date of first study treatment administration to the date of first documented tumor progression or death due to any cause, whichever occurs first.
Duration of response (DOR) | from the first drug administration up to two years
  Time from first documented response (CR or PR) until documented disease progression or death, whichever occurs first.
Disease Control Rate (DCR) | from the first drug administration up to two years
  Proportion of patients whose best overall response is either CR, PR, or SD according to RECIST v1.1.
Overall survival (OS) | from the first drug administration up to two years
  Time from the date of first study treatment administration to the date of death due to any cause.
Safety and tolerability | up to 90 days after last study treatment administration
  Incidence of Adverse Event reported per CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Xin Huang, Principal Investigator — Sun Yat-sen University Cancer Centre
Locations (1):
- Sun Yat-sen University Cancer Centre, Guangzhou, Guangdong, China